CLINICAL TRIAL: NCT02325128
Title: Augmentation of Exposure Therapy for High Levels of Social Anxiety Using Post-exposure Naps
Acronym: SANAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Edward F. Pace-Schott, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2014P001501/MGH
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Social Anxiety Disorder; Sleep Laboratory
Keywords: social anxiety; exposure therapy; extinction; sleep-dependent memory consolidation
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Post-Exposure Nap (Experimental): Sleep-enhancement of extinction memory: At the end of the third and fourth of 5 exposure therapy sessions, all participants deliver a speech designed to elicit significant social anxiety. Following this speech, this arm will be given a 2-hour sleep opportunity with polysomnographic (PSG) monitoring.
  Interventions: Behavioral: Sleep-enhancement of extinction memory
- Post-Exposure Wake (Active Comparator): At the end of the third and fourth of 5 exposure therapy sessions, all participants deliver a speech designed to elicit significant social anxiety. Following this speech, this arm will be instrumented for PSG but, instead of napping, will undergo 2 hours of quiet wakefulness. Therefore, this arm will not undergo sleep-enhancement of extinction memory.
  Interventions: Behavioral: Sleep-enhancement of extinction memory

INTERVENTIONS:
Behavioral: Sleep-enhancement of extinction memory — Recent reports show that sleep promotes memory consolidation. The investigators' preliminary findings suggest sleep may enhance the therapeutic extinction memories acquired during exposure therapy. For sleep-enhancement of extinction memory, the current intervention uses post-exposure naps as a means to provide sleep in close temporal proximity to the encoding of memory for the extinction social exposure fears in individuals with severe social anxiety symptoms.

SUMMARY:
Investigators will examine whether post-exposure naps can be used to strengthen therapeutic extinction memories formed during exposure therapy for extreme social anxiety. Thirty-two individuals with high levels of social anxiety, evidenced by scores of 60 or greater on the Liebowitz Social Anxiety Scale, by self-report during a clinical interview and by demonstrated enhanced psychophysiological reactivity when imagining a socially stressful scenario, will be enrolled as one of four participants in one of eight successive offerings of a validated 5-session exposure-based group treatment for extreme social anxiety. The third and fourth sessions conclude with each participant delivering a speech on a topic individually chosen to elicit significant social anxiety. Following these sessions, participants will go to the sleep laboratory where two will be given a 2-hour sleep opportunity with polysomnographic (PSG) monitoring and two will be similarly instrumented but undergo 2 hours of monitored quiet wakefulness. Before and after treatment, participants will be individually assessed for social anxiety symptoms using standardized self-report instruments and a Trier Social Stress Test (TSST) modified for continuous psychophysiological monitoring. Ambulatory monitoring of home sleep will also be obtained using actigraphy and sleep diaries. The investigators hypothesize that, post treatment, those individuals who napped will show greater questionnaire-based clinical improvement as well as lesser psychophysiological reactivity during the modified TSST compared to those who remained quietly awake. The investigators further hypothesize that characteristics of sleep quality and architecture during naps, specifically durations of total sleep, REM and slow-wave sleep, as well as REM continuity, will predict greater clinical improvement and lesser psychophysiological reactivity to the TSST in those who napped following their third and fourth therapy sessions. Positive results will provide the first proof-of-principle for sleep augmentation of exposure therapy for clinically significant extreme social anxiety.

DETAILED DESCRIPTION:
Widely replicated studies demonstrate that sleep can enhance memory consolidation. Potential clinical applications of such findings have only begun to be explored. The investigators have recently shown that nocturnal sleep following simulated exposure therapy for high levels of spider fear reduced both psychophysiological and self-reported reactivity when participants were re-exposed to the same and to novel spider stimuli. The proposed research will extend these findings to the more debilitating and clinically important condition of extreme social anxiety. The investigators will examine whether post-exposure naps can be used to strengthen therapeutic extinction memories formed during exposure exercises used in the behavioral treatment of extreme social anxiety. A total of 32 individuals with high levels of social anxiety, evidenced by scores of 60 or greater on the Liebowitz Social Anxiety Scale, self-report during a clinical interview and demonstrated enhanced psychophysiological reactivity when imagining a socially stressful scenario, will be enrolled in an exposure-based group treatment for extreme social anxiety. Eight successive therapy groups of 4 patients each will be offered during the 2-year funding period. The third and fourth sessions of this validated 5-week/5-session treatment will involve each participant delivering a speech on a topic individually chosen to elicit significant social anxiety. Following both of these sessions, all 4 participants will go to the nearby Massachusetts General Hospital sleep laboratory where 2 will be given a 2-hour sleep opportunity with polysomnographic (PSG) monitoring and the other 2 will be similarly instrumented but undergo 2 hours of monitored quiet wakefulness (prior to session 3 participants will be randomized to the sleep or wakefulness arm). Before beginning treatment and within several days following the final treatment session, all participants will be individually assessed for social anxiety symptoms using standardized self-report instruments. At these same times, they will undergo a Trier Social Stress Test (TSST) modified for continuous psychophysiological monitoring that also includes repeated Subjective Units of Distress (SUDS) self report and sampling for salivary cortisol. In addition to laboratory PSG, ambulatory monitoring of home sleep with actigraphy and sleep diaries will take place at pre-treatment baseline and during the last 3 weeks of treatment. The investigators hypothesize that those individuals allowed a 2-hour sleep opportunity following exposure sessions, compared to those who remained quietly awake, will show greater questionnaire-based clinical improvement as well as lesser psychophysiological and SUDS reactivity during the modified TSST. The investigators further hypothesize that characteristics of sleep quality and architecture during naps, specifically durations of total sleep, REM sleep and slow-wave sleep as well as REM continuity, will predict clinical improvement and diminished TSST reactivity in those who napped. To help ensure that observed sleep effects are attributable to the two 2-hour sleep opportunities, the investigators will control for actigraph and diary-measured sleep quality during treatment. Positive results will provide the first proof-of-principle for sleep augmentation of exposure therapy for a clinically significant extreme social anxiety.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. Treatment-seeking individuals diagnosed with Social Anxiety Disorder using the Structured Clinical Interview for DSM-IV56 (DSM-5 SCID once available)
2. A score > 60 on the Liebowitz Social Anxiety Scale (LSAS)13
3. 18-40 years of age
4. Proficient in English
5. Normal or corrected to normal vision
6. Able to give informed consent
7. Willingness and ability to comply with the requirements of the study protocol
8. Meets psychophysiological screening criteria for inclusion carried out as follows:

   * During a 5-min. baseline period, the candidate participant will sit quietly with skin conductance and orbicularis oculi EMG levels being recorded.
   * Toward the end of this period a loud acoustic stimulus will be presented several times and blink startle EMG and SCR will be recorded.
   * The candidate subject will then be asked to describe, for 2 min., their most fearful and upsetting past social experience.
   * They will then be instructed to silently reimagine this experience as vividly as possible.
   * During this imagination period, the loud acoustic stimulus will again be presented several times and blink startle EMG and SCR will be recorded.
   * Participants for whom mean SCR and blink startle EMG during the imagining period measurably exceed the means of these measures during baseline will be retained in the study whereas those for whom these measures do not change or are reduced will be excluded.
   * This procedure will help ensure that those included in the study will show potentiation of physiological reactivity while anticipating exposure to public speaking.

Exclusion Criteria:

1. Any potentially confounding medical illness
2. Lifetime history of any neurological illness or injury including neurodegenerative disorders or dementia, stroke, seizure disorders, neurosurgical procedures, head injury resulting in loss of consciousness for greater than 5 min.
3. Lifetime history, diagnosed by DSM-IV criteria (or DSM-5 once its SCID available), of bipolar disorder, schizophrenia or other psychotic disorder, pervasive developmental disorder, chronic mental disorder due to a medical condition or other potentially confounding chronic mental disorder.
4. Current major depressive, dysthymic or anxiety disorder other than Social Anxiety Disorder or other potentially confounding current mental disorder diagnosed by DSM-IV criteria (or DSM-5 once its SCID available).
5. DSM-IV substance abuse or dependence within the last year, lifetime history of hospitalization for substance abuse (determined at clinical interview) or positive urine toxicology screen at the time of the clinical interview
6. Any evidence of suicidal ideation, violent behavior or psychosis at the clinical interview
7. Use of psychiatric medication within 4 weeks of study (with the exception of 6 weeks for fluoxetine)
8. Current psychotherapy for Social Anxiety Disorder
9. Any indication of a sleep disorder, particularly sleep-disordered breathing, on the Pittsburgh Structured Clinical Interview for Sleep Disorders
10. Sleep onset latency > 1 hr, total sleep time < 5 hr or typical bed time later than 3 AM
11. Overnight shift work or recent travel across multiple time zones
12. > 4 caffeinated beverages per day or > 11 alcoholic beverages per week
13. Nicotine use

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Leibowitz Social Anxiety Scale | 5 weeks
  Validated self-report scale used to assess degree of social anxiety
Fear-potentiated startle | 5 weeks
  Orbicularis oculi electromyography used to record the blink startle response to loud tones while anticipating delivering a speech to an audience and during an initial baseline period; difference measure obtained by subtracting the baseline startle response from the startle response recorded while anticipating a fearful situation

SECONDARY OUTCOMES:
Fear of Negative Evaluation Scale | 5 weeks
  Validated self-report scale to assess fear of negative evaluation by others
Social Phobia and Anxiety Inventory | 5 weeks
  Validated self-report scale to assess degree of social anxiety
Clinical Global Impressions Scale | 5 weeks
  Validated clinician-based evaluation of symptom severity and impairment of functioning
Pre- to-post TSST change in Spielberger State-Trait Anxiety Inventory-State portion score | up to 5 weeks
  Validated self-report scale to assess an individual's current level of anxiety; administered before and after TSST; pre-post difference indexes degree to which the TSST increased state anxiety
Subjective Units of Distress Ratings | 5 weeks
  Validated, individually anchored, rating of subjective distress on a scale of 0 to 100
Pre- to-post TSST change in salivary cortisol | up to 5 weeks
  Salimetrics oral swab used to collect and analyze salivary cortisol levels at baseline and at time points reflective of maximum levels evoked by the speech-performance phase of the TSST.
Fear potentiation of loud-tone evoked heart-rate acceleration (HRA) and skin conductance response (SCR) | 5 weeks
  Electrocardiography records HRA and electrodermal measures record SCR evoked by loud tones while anticipating delivering a speech to an audience; responses to same stimuli recorded during an initial baseline period; difference measure obtained by subtracting baseline HRA and SCR from HRA and SCR recorded while anticipating a fearful situation.
Increase in baseline heart rate from baseline to performance phases of TSST | up to 5 weeks
  Electrocardiography records maximum heart rate during an initial baseline; difference measure subtracts baseline from the maximum heart-rate during actual delivery of the speech in TSST performance phase.
Increase in mean corrugator supercilii EMG from baseline to performance phases of TSST | 5 weeks
  Electromyography records mean corrugator supercilii muscle tone during baseline period; difference measure subtracts baseline from the mean corrugator supercilii muscle tone recorded during actual delivery of speech in the TSST performance phase.

OTHER OUTCOMES:
NEO-PI-R Neuroticism and Extraversion total scores | 5 weeks
  Validated and widely used scale to quantify dimensions of personality hypothesized by the 5-factor model; only Neuroticism and Extraversion factors evaluated
Social Avoidance and Distress Scale | 5 weeks
  Validated scale used to assess the degree of avoidance of social situations
Social Probability and Social Cost Questionnaire | 5 weeks
  Validated instrument to assess degree to which an individual anticipates the likelihood and severity of harm resulting from social encounters
Pre- to-post TSST change in Positive and Negative Affect Scale subtotals | up to 5 weeks
  Validated self-report scale to assess participants' current level of positive and negative emotions; administered before and after the TSST; pre-post differences index degree to which the TSST decreased levels of positive emotion and increased levels of negative emotion
Pre- to-post TSST change in Stanford Sleepiness Scale subtotals | up to 5 weeks
  Validated self-report scale to assess current level of sleepiness; administered before and after the TSST; pre-post differences index the degree to which the TSST increased subjective arousal (inverse of self-reported sleepiness)
Rate and number of spontaneous SCRs during baseline, preparation and performance phases of TSST | 5 weeks
  SCR measures sympathetic nervous system (SNS) activation. Spontaneous SCRs index the degree to which the SNS is phasically activated. A difference measure is obtained between the rate of spontaneous SCRs during baseline phase and rate during the speech preparation and performance phases of the TSST.
Rate of mean HR decline from performance to late recovery phases of the TSST | 5 weeks
  Decline in HR from an anticipated maximum during actual performance of the speech until the end of both recovery phases (early and late) following speech; indexes degree to which participant able to self-soothe following stressor
Social Interaction Self-Statements Test | 5 weeks
  Self-report test to assess participants' self evaluation following a specific social encounter given at the end of both TSSTs.

CONTACTS AND LOCATIONS:
Overall Officials: Edward F Pace-Schott, Ph.D., Principal Investigator — Massachusetts General Hospital and Harvard Medical School
Locations (2):
- United States (2):
  - Massachusetts General Hospital, One Bowdoin Square, Boston, Massachusetts
  - Massachusetts General Hospital-East, Building 149, Charlestown, Massachusetts

REFERENCES:
- [Background] Pace-Schott EF, Verga PW, Bennett TS, Spencer RM. Sleep promotes consolidation and generalization of extinction learning in simulated exposure therapy for spider fear. J Psychiatr Res. 2012 Aug;46(8):1036-44. doi: 10.1016/j.jpsychires.2012.04.015. Epub 2012 May 10. PMID 22578824
- [Background] Zalta AK, Dowd S, Rosenfield D, Smits JA, Otto MW, Simon NM, Meuret AE, Marques L, Hofmann SG, Pollack MH. Sleep quality predicts treatment outcome in CBT for social anxiety disorder. Depress Anxiety. 2013 Nov;30(11):1114-20. doi: 10.1002/da.22170. Epub 2013 Aug 26. PMID 24038728
- [Result] Pace-Schott EF, Bottary RM, Kim SY, Rosencrans PL, Vijayakumar S, Orr SP, Lasko NB, Goetter EM, Baker AW, Bianchi MT, Gannon K, Hoeppner SS, Hofmann SG, Simon NM. Effects of post-exposure naps on exposure therapy for social anxiety. Psychiatry Res. 2018 Dec;270:523-530. doi: 10.1016/j.psychres.2018.10.015. Epub 2018 Oct 9. PMID 30340182